CLINICAL TRIAL: NCT06060353
Title: A Pragmatic Randomized Controlled Trial of Regulation-Focused Psychotherapy (RFP-C) for Children With Externalizing Problems
Brief Title: Randomized Controlled Trial of Regulation-Focused Psychotherapy (RFP-C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Center for Regulation Focused Psychotherapy (Unknown)
Responsible Party: Principal Investigator, Sibel Halfon, Associate Professor, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFP-C
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Childhood Externalizing Disorder; Childhood Oppositional Defiant Disorder; Childhood Conduct Disorder
Keywords: Regulation Focused Psychotherapy; Implicit Emotion Regulation; Externalizing Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regulation Focused Psychotherapy (RFP-C) (Experimental)
  Interventions: Behavioral: Regulation Focused Psychotherapy (RFP-C)
- Parental Awareness and Child Social Skills Group (Active Comparator)
  Interventions: Behavioral: Parental Awareness and Child Social Skills Group

INTERVENTIONS:
Behavioral: Regulation Focused Psychotherapy (RFP-C) — Regulation-focused psychotherapy for children (RFP-C; Hoffman, Rice, & Prout, 2016) is a manualized, psychodynamic play therapy. Through 20 sessions (16 with the child and four parent meetings), RFP-C allows the child to understand the ways distressing affects are avoided and to explore alternative ways of coping with unpleasant affect. The clinician works to increase the child's understanding that all behavior, especially oppositional and disruptive behavior, has meaning in the service of emotional and behavioral regulation. This work is also done with the parents to better support the child in achieving symptom reduction and increased emotion regulation.
  Arms: Regulation Focused Psychotherapy (RFP-C)
Behavioral: Parental Awareness and Child Social Skills Group — Parental awareness and child social skills group is a manualized group psychotherapy that involves twelve parallel sessions conducted separately with parents and children. The parent group involves modules related to psycho-education, role-play and awareness building activities on child needs & rights, child temperament, praise & acceptance, child play, limit setting, anger management, transmission of parenting styles through genograms and family trees. With children, the groups involve psycho-education and play based activities to build awareness on children's rights, temperament, feelings, play & relationship skills, empathy & praise, anger management.
  Arms: Parental Awareness and Child Social Skills Group

SUMMARY:
Regulation Focused Psychotherapy for Children (RFP-C) is a manualized, time-limited psychodynamic treatment for children with externalizing symptoms. RFP-C also holds the potential to treat a wider range of psychopathology, including comorbid internalizing conditions, because it aims to improve emotion regulation which is a transdiagnostic component of childhood mental health. This study will replicate previous findings supporting the efficacy of RFP-C. It will test the effectiveness of RFP-C in parallel groups via a pragmatic Randomized Controlled Trial (RCT) conducted at Istanbul Bilgi University's outpatient clinic in Istanbul, Turkey with a sample of 80 children with externalizing and comorbid internalizing/externalizing problems in comparison to a parental awareness and child social skills group. Primary outcomes will be child externalizing problems and oppositional defiance problems. The treatment's effectiveness and change mechanisms will be investigated both at the end of treatment (primary endpoint) and at 6-month follow-up (secondary endpoint). The project results will provide preliminary answers about the active ingredients of RFP-C, help improve therapeutic interventions, and design optimal treatments for externalizing problems.

ELIGIBILITY:
Inclusion Criteria:

1. Children must be between the ages of 6-12 years of age
2. Meet criteria for clinical levels of externalizing problems on the SDQ
3. Parent(s) able to attend four sessions of parent meetings

Exclusion Criteria:

1. Solely emotional problems and non-clinical problem levels (as assessed by the SDQ)
2. Primary diagnosis of psychosis or eating disorders (as assessed by KSADS-PL)
3. Risk for suicide and/or severe violence risk (as assessed by KSADS-PL)
4. Current enrollment in another psychosocial treatment
5. Intellectual disability or major developmental delay (e.g. moderate/severe autism spectrum disorder) (as assessed by KSADS-PL & WASI)
6. Families with high risk of domestic abuse
7. Parents with acute psychosis (as assessed by SCID)
8. Parents with severe substance abuse and dependence (as assessed by SCID)
9. Parents with intellectual disability (as assessed by WASI)
10. Parents with acute risk of harm to self and others (as assessed by SCID)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Strengths and Difficulties Questionnaire - Parent version (SDQ-P; Goodman, 2001) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Strengths and Difficulties Questionnaire - Parent version (SDQ-P; Goodman, 2001) is a 25-item scale that asks parents to rate their children's emotional and behavioral difficulties on a 3-point Likert scale, ranging from 0 = not true to 2 = very true. The questionnaire is composed of five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity-Inattention, Peer Problems and Prosocial. In addition, the SDQ-P yields Internalizing Difficulties, Externalizing Difficulties and Total Difficulties scale scores. SDQ-P was demonstrated to be a valid and reliable scale for use in Turkish children and adolescents (Yalın et al., 2013).
Turgay DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) Disruptive Behavior Disorders Rating Scale (T-DSM-IV-S; Turgay, 1994) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Turgay DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) Disruptive Behavior Disorders Rating Scale (T-DSM-IV-S; Turgay, 1994) is based on DSM-IV diagnostic criteria and examines hyperactivity/impulsivity, inattention, opposition-defiance, and conduct disorder. Symptoms are scored on a four-point Likert scale (0= not at all, 1= just a little, 2= quite a bit, and 3= very much). T-DSM-IV-S has shown good reliability and validity.

SECONDARY OUTCOMES:
Me and My Feelings Questionnaire (M&MF; Deighton et al., 2013) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Me and My Feelings Questionnaire (M&MF; Deighton et al., 2013) is a child-report measure consisting of total short 16-items: 10-items of emotional difficulties scale and 6-items of behavioral difficulties scale. It is scored on a 3-point likert scale (0 = "never expressed", 1 = "sometimes expressed", 2 = "always expressed"). Total score of scales are calculated as the sum of item scores with threshold values 10 for the emotional difficulties and six for the behavioral difficulties. Higher scores of each set of difficulties indicate the probability of mental health problems. The scale has been adapted to Turkish with good reliability and validity (İlnem, 2020).
Emotion Regulation Checklist (ERC; Shields & Cicchetti, 1997) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Emotion Regulation Checklist (ERC; Shields & Cicchetti, 1997) is a parent-report measure of children's emotion regulation characteristics and involves 24-items rated on a 5-point likert scale (1 = "never" to 5 = "always"). It taps into two factors one of which is emotional lability and negativity defined as arousal, anger dysregulation, and mood changes; and the second is emotion regulation defined as socially appropriate emotional displays, empathy, and emotional selfawareness. The scale has been adapted to Turkish with good reliability and validity (Batum & Yagmurlu, 2007).
The Emotion Awareness Questionnaire (EAQ-30; Rieffe et al., 2008) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  The Emotion Awareness Questionnaire (EAQ-30; Rieffe et al., 2008) aims to identify how children and adolescents feel and think about their feelings. The EAQ (30 items) was designed with a six-factor structure describing six aspects of emotional functioning: (1) Differentiating Emotions, (2) Verbal Sharing of Emotions, (3) Not Hiding Emotions (formerly Acting Out), (4) Bodily Awareness of Emotions, (5) Attending to Others' Emotions, and (6) Analyses of Emotions. Respondents are asked to rate the degree to which each item is true about them on a three-point scale (1 = not true, 2 = sometimes true, 3 = often true). The scale has been adapted to Turkish with good reliability and validity (İnceman, 2017).
The Children's Global Assessment Scale (CGAS; Schaffer et al., 1983) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2)
  The Children's Global Assessment Scale (CGAS; Schaffer et al., 1983) is a numeric scale (from 1 to 100) used by mental health clinicians to rate the global functioning of children under the age of 18 on a scale of 0 to 100. 90- 81 range is scored when there is "good functioning in all areas; security in family, school, and with peers with only transient difficulties and everyday worries"; 50-41, when there is "moderate degree of interference in functioning in most social areas or severe impairment of functioning in one area"; and 20-11, when there is "need for considerable supervision to prevent hurting others or self or to maintain personal hygiene or gross impairment in all forms of communication". The scale has been adapted to Turkish with good reliability and validity (Gökler et al., 2004).
Parental Stress Index - Short Form (PSI-SF; Abidin, 1983) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Parental Stress Index - Short Form (PSI-SF; Abidin, 1983) is a 36-item parent-report scale.The PSI-SF contains 36 items divided into three subscales, each composed of 12 items: "Parental distress"; "Parent-child dysfunctional interaction"; "Difficult child". Each item is rated on a 5-point likert scale from 1 = "strongly disagree" to 5 = strongly agree". The PSI-SF gives three subscores and a total distress score. The scale has been adapted to Turkish with good reliability and validity (Ertan et al., 2008).
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2), 36th week (T3)
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) is an instrument measuring emotion regulation problems in adults (to be used with parents in the current study). The scale comprises 36 items that are rated on a 5- point likert scale from 1 = "almost never" to 5 = "almost always", with higher scores indicating a difficulty of emotion regulation. The scale produces scores on the following subscales: (a) lack of awareness of emotional responses; (b) lack of clarity of emotional responses; (c) nonacceptance of emotional responses; (d) limited access to effective strategies; (e) difficulties in controlling impulsive behavior when experiencing negative affect; and (f) difficulties in engaging goal directed behavior when experiencing negative affect as well as a total disregulation score. The scale has been adapted to Turkish with good reliability and validity (Yiğit & Güzey-Yiğit, 2017).

OTHER OUTCOMES:
Adverse Childhood Experiences Scale (ACE; Dube et al., 2004) | Time Frame: Baseline (T0)
  Adverse Childhood Experiences Scale (ACE; Dube et al., 2004) is a parent-report scale to assess retrospectively forms of abuse, neglect, and household dysfunction (i.e., witnessing domestic violence, separation and mental illness in the family) in the current study. Scores range from 0-10 on the ACE, with the latter representing full exposure at some point in the first 18 years of life, to all forms of household dysfunction and abuse detailed in the questionnaire.It has a parent and a child version. The scale has been adapted to Turkish by Gunduz et al. (2018).
The Therapeutic Alliance Scale for Children-revised (TASC-r; Creed &Kendall, 2005) | Time Frame: Baseline (T0), Mid-Treatment (T1), End of Treatment (T2)
  The Therapeutic Alliance Scale for Children-revised (TASC-r; Creed &Kendall, 2005) is a 12-item tool that measures alliance across the three dimensions of task, bond and goals and covers both positive and negative aspects of therapeutic alliance. Each response is rated on a four point Likert scale (i.e. ''not at all like my client'' to ''very much like my client''). It has been found to have adequate reliability and validity in Turkey (Bulut, et al., 2023).
Wechsler Abbreviated Scale of Intelligence (WASI-II; Weschler, 1999) | Time Frame: Baseline (T0)
  Wechsler Abbreviated Scale of Intelligence (WASI-II; Weschler, 1999) is a brief measure of verbal and nonverbal intelligence administered by trained researchers to parents and children.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffman, L., Rice, T., & Prout, T. (2015). Manual of Regulation-Focused Psychotherapy for Children (RFP-C) with externalizing behaviors: A psychodynamic approach. Routledge.